CLINICAL TRIAL: NCT01533363
Title: Patient Comfort After Stapled Hemorrhoidopexy Long Term Results of a Randomized Controlled Trial
Brief Title: Study About Patient Comfort and Long-term Outcome After Stapled Hemorrhoidopexy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Asad Kutup, Senior Surgeon, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1612
Record Dates: First submitted 2012-02-05; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Internal Hemorrhoids
Keywords: Hemorrhoids; Surgery; Hemorrhoidopexy; Milligan Morgan
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stapled hemorrhoidopexy (Active Comparator): surgical procedure to treat hemorrhoids
  Interventions: Procedure: Stapled hemorrhoidopexy
- Milligan Morgan (Active Comparator): surgical procedure to treat hemorrhoids
  Interventions: Procedure: Milligan Morgan

INTERVENTIONS:
Procedure: Stapled hemorrhoidopexy
  Other Names: Ethicon PPH 01
  Arms: Stapled hemorrhoidopexy
Procedure: Milligan Morgan
  Arms: Milligan Morgan

SUMMARY:
The purpose of this study was to determine the influence on Patient comfort after Stapled Hemorrhoidopexy versus Milligan Morgan (two surgical procedures)in third degree circular hemorrhoids.

DETAILED DESCRIPTION:
There are well known advantages in the short-outcome, however, there are still some uncertainties about the long-term results and recurrence rates, and only a few data of randomized trials are available.

In most studies the patient population was heterogeneous with a varied degree of treated hemorrhoids, and different surgical procedures were performed. Therefore we initiated this prospective randomized controlled study of a homogeneous patient population with only circular third-degree hemorrhoids and clearly defined operative procedures. All patients with symptomatic, reducible circular third-degree hemorrhoidal disease were randomly assigned to undergo either the Milligan-Morgan technique or the stapling procedure. Patients were excluded from the study if they had single third-degree hemorrhoids, acute incarcerated hemorrhoids, intercurrent acute anal fissure and/or acute anal fistula, or prior hemorrhoidectomy. The main end point parameter of this study was to compare both groups with respect to patient comfort and postoperative pain. Secondary end points included the long-term recurrence rate of hemorrhoidal disease after a minimum of 4 years.

ELIGIBILITY:
Inclusion Criteria:

* third degree circular hemorrhoids
* symptomatic
* reducible

Exclusion Criteria:

* single third-degree hemorrhoids
* acute incarcerated hemorrhoids
* intercurrent acute anal fissure
* acute anal fistula
* prior hemorrhoidectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2000-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | within the first 30 days after surgery

SECONDARY OUTCOMES:
long-term recurrence rate | up to 5 years after surgery
  Secondary end points included the long-term recurrence rate of hemorrhoidal disease after a minimum of 4 years. Postoperative morbidity such as bleeding, wound infection, urinary retention, and itching and burning, and transient incontinence symptoms, and parameters such as length of hospital stay and operating time were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Jakob R Izbicki, MD, Study Chair — Dept. of Surgery, Martinistreet 52, University Hospital Hamburg Eppendorf, 20246 Hamburg

REFERENCES:
- [Background] Gravie JF, Lehur PA, Huten N, Papillon M, Fantoli M, Descottes B, Pessaux P, Arnaud JP. Stapled hemorrhoidopexy versus milligan-morgan hemorrhoidectomy: a prospective, randomized, multicenter trial with 2-year postoperative follow up. Ann Surg. 2005 Jul;242(1):29-35. doi: 10.1097/01.sla.0000169570.64579.31. PMID 15973098